CLINICAL TRIAL: NCT06484673
Title: Randomized, Two-way, Two-period, Single Oral Dose, Open-label, Crossover, Bioequivalence Study to Compare Bosentan 32 mg Dispersible Tablets Versus Tracleer® 32 mg Tablets for Oral Suspension (Tracleer® 32 mg Dispersible Tablet) (Bosentan), in Healthy Subjects Under Fasting Condition
Brief Title: Bioequivalence Study to Compare Bosentan 32 mg Dispersible Tablets Versus Tracleer® 32 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1293-2024
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bosentan 32 mg Dispersible Tablets (Experimental): Bosentan 32 mg Dispersible Tablets
  Interventions: Drug: Bosentan Dispersible Tablets; Drug: Tracleer Tablet for Oral Suspension
- Tracleer® 32 mg Tablets for Oral Suspension (Active Comparator): Tracleer® 32 mg Tablets for Oral Suspension (Tracleer® 32 mg Dispersible Tablet) (Bosentan)
  Interventions: Drug: Bosentan Dispersible Tablets; Drug: Tracleer Tablet for Oral Suspension

INTERVENTIONS:
Drug: Bosentan Dispersible Tablets — 1 tablet of 32 mg Bosentan
Drug: Tracleer Tablet for Oral Suspension — 1 tablet of 32 mg Bosentan

SUMMARY:
Randomized, two-way, two-period, single oral dose, open-label, crossover, bioequivalence study to compare Bosentan 32 mg Dispersible Tablets versus Tracleer® 32 mg Tablets for Oral Suspension (Tracleer® 32 mg Dispersible Tablet) (Bosentan), in healthy subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male & aged between eighteen to forty-five years (18 - 45), both inclusive.
* The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
* The results of medical history, physical examination, vital signs & conducted medical laboratory tests are normal as determined by the clinical investigator.
* The subject tested negative for Hepatitis B (HBsAg), Hepatitis C (HCVAb) and human immunodeficiency virus (HIVAb).
* There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* The subject has normal cardiovascular system, pulmonary system & ECG recording.
* The subject kidney and liver functions (AST & ALT enzymes) tests are within normal range.
* The subject blood pressure is ≥ 110/70 mmHg before dosing.

Exclusion Criteria:

* The subject is a heavy smoker (more than 10 cigarettes per day).
* The subject has suffered an acute illness one week before dosing.
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is vegetarian.
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 48 hours after dosing in both study periods.
* The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.
* The subject has consumed any drugs that may affect pharmacological or pharmacokinetic properties of Bosentan. (for example: fluconazole, amiodarone, ketoconazole, itraconazole, amprenavir, erythromycin, fluconazole, diltiazem, Cyclosporine A, Glyburide, Norethindron, Ethinyl estradiol, Simvastatin, lopinavir, ritonavir, Rifampin) two weeks before and after the study and during the study.
* The subject suffer from phenylketonuria disorder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Maximum concentration obtained (Cmax) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data Cmax
AUC from time 0 to last collection time t (AUC0-t) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data AUC0-t

SECONDARY OUTCOMES:
AUC from time 0 to infinity (AUC0-inf) | 23 hours
  Description Statistics
Time of the maximum measured plasma concentration (Tmax) | 23 hours
  Description Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- ACDIMA Biocenter, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No